CLINICAL TRIAL: NCT06161779
Title: Sun Yat-sen Memorial Hospital, Sun Yat-sen University
Brief Title: Submental Flap for the Reconstruction of Hypopharyngectomy
Acronym: SMFRLPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-123-01
Record Dates: First submitted 2023-09-04; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Head and Neck Cancers - Hypopharyngeal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Submental artery flap reconstruction group (Experimental)
  Interventions: Other: Surgical reconstruction

INTERVENTIONS:
Other: Surgical reconstruction — submental artery island flap (SMAIF) for the reconstruction of laryngeal and hypopharyngal defects after the surgical resection of hypopharyngeal cancer

SUMMARY:
The goal of this observational study is to assess the safety and efficacy of submental artery island flap (SMAIF) in the reconstruction of laryngeal and hypopharyngal defects after the surgical resection of hypopharyngeal cancer. The main questions it aims to answer are:

* The survival of SMAIF and the recovery of laryngeal function.
* The oncologic outcomes of SMAIF comparing with other reconstructions or radiotherapy.

Participants will underwent partial laryngectomy and hypopharyngectomy and reconstruction of SMAIF. Postoperative adjuvant radiotherapy will be recommented when adverse pathologic features were noted.

DETAILED DESCRIPTION:
1. Introduction:

   Hypopharyngeal cancer is a common malignant tumor of the head and neck, ranking 27th in the world in 2020. Current treatments for hypopharyngeal carcinoma include surgical resection plus postoperative adjuvant radiotherapy (SRT) and concurrent radiochemotherapy (CRT). Hypopharyngeal cancer often invades the larynx, and both surgery and radiotherapy can cause laryngeal insufficiency and affect the quality of life of patients. Repair of laryngeal and hypopharyngeal defects after surgical resection of hypopharyngeal carcinoma includes pull-in suture, adjacent tissue flap or free flap repair. The submental artery island flap (SMAIF) is located in the same surgical field as hypopharyngeal carcinoma resection, and the thickness of the flap is suitable, which has the advantages of convenient harvest, stable blood supply and high accessibility. The SMAIF was used to repair the hypopharynx, but the laryngeal defeat was ignored. This study is a prospective single-arm study, which is aimed to assess the safety and efficacy of SMAIF to repair the laryngeal and hypopharyngeal defects of the resection of T2-T3 hypopharyngeal carcinoma. The oncological results and laryngeal function parameters will be recorded. The ultimate gold of the study is to obtain a simple and effective reconstruction method for locally advanced hypopharyngeal cancer.
2. Background:

   Hypopharyngeal squamous cell cancer (HPSCC) is a common head and neck malignant tumor, ranking 27th among new malignant tumors in the world in 2020 [1]. HPSCC has an insidious onset, is prone to submucosal infiltration and growth, and cervical lymph node metastasis occurs in the early stage. When discovered, most are in the late stage, and have the worst prognosis among head and neck squamous cell carcinomas. Surgery plus postoperative radiotherapy (SRT) or radical concurrent chemoradiotherapy (CRT) is the mainstream treatment for HPSCC [2]. The 5-year overall survival rate of the SRT group was 44.6%, while that of the CRT group was 40.4%. SRT has a better 5-year survival rate than CRT (HR=0.89) [3]. HPSCC often invades the larynx. Regardless of surgery or radiotherapy, it can cause cricoarytenoid joint impairment, laryngeal cartilage necrosis and other laryngeal injuries after treatment, followed by dyspnea, dysphagia and other laryngeal insufficiency, which requires long-term tracheotomy or with a gastric tube affects the patient's quality of life.

   Of the SRT group, due to the different proportions of total laryngectomy and different repair methods among different hospitals, the laryngeal function preservation rate among the SRT groups varies greatly [3]. Among them, Jang et al. reported the largest surgical sample size (n=177), with a higher proportion of larynx-preserving surgery. The reported larynx-preserving rate (LPR) after hypopharyngeal cancer surgery was about 60%, but it was still inferior to the 76.6% of CRT [4]. The inclusion criteria of Jang and others are relatively consistent with the preset inclusion conditions of this clinical trial, so we selected Jang's LPR as the baseline. Reconstruction of laryngeal and hypopharyngeal defects after surgical resection of HPSCC include pulling-in suture, adjacent tissue flap or free skin flap repair [5]. T3 hypopharyngeal cancer cases often invade the ipsilateral paraglottic space and require resection of the ipsilateral hemi-larynx. Therefore, simultaneous repair of hemi-laryngeal defect and hypopharyngeal defect remain a challenge for the surgeons.

   In the early stage, we used adjacent platysma muscle flap transfer to repair defects of the larynx and hypopharynx, and achieved satisfactory results [6]. However, the platysma flap has no definite perforating arteries and the size of the donor is limited. At the same time, the platysma flap tissue volume is small, making it difficult for the hypopharyngeal piriform sinus to reach normal size after repair. We also used the radial forearm perforator flap (RFPF) to repair posterior pharyngeal wall defects during resection of HPSCC [7]. However, free flaps require microvascular anastomosis, which is technically difficult, risky, and time-consuming. It often requires two groups of surgeons, tumor resection and reconstruction, to perform the surgery at the same time. These factors also limit the use of free flaps for repair after hypopharyngeal cancer resection.

   The submental artery island flap (SMAIF), referred to as the submental flap, is an axial flap that is located in the same surgical field as hypopharyngeal cancer resection. The thickness of the flap is moderate and suitable for the hypopharynx, and it has the advantages of easy harvest, stable blood supply, and high accessibility [8]. Ye et al. studied 27 cases of submental flap for the postoperative defect repair of pharyngeal SCC. One case (3.7%) occurred flap necrosis; meanwhile, no metastasis of lymph node biopsy in cervical area I [9], suggesting that SMAIF is safe and applicable as a donor. However, in this study, the submental flap only repaired the hypopharyngeal defect, and the laryngeal defect was ignored.

   We have performed 3 cases of SMAIF repair in T3 HPSCC. The conventional donor area of 6cm × 8cm skin island is sufficient to cover the defect of ipsilateral larynx and pyriform sinus. No case of skin flap ischemic necrosis occurred. The nasogastric tube can be successfully removed at postoperative 2 to 4 weeks and the patient can eat orally. Therefore, we plan to conduct a prospective single-arm study of SMAIF repair of laryngeal and hypopharyngeal defects after HPSCC resection, and observe the oncological results and postoperative laryngeal function including respiratory, swallowing, and voice function, and compared with historical series of HPSCC treated with SRT or CRT, to explore the safety and effectiveness of this flap for repairing laryngeal and hypopharyngeal defects. In order to obtain a reconstruction technique with a good accessibility, safety and effectiveness for the surgical treatment of locally advanced HPSCC.
3. Study Design:

   This study is a single-armed observational study aimed to investigate the role of submental flap on the preservation of laryngeal function after surgical resection of HPSCC. The study duration is 5 years, and 40 patients with HPSCC will be enrolled.
4. Intervention:

   4.1 After patients with hypopharyngeal cancer are admitted to the hospital, the primary site and clinical stage of the tumor will be determined based on imaging and pathological examinations such as laryngoscopy, magnetic resonance (MR) or CT, and those who meet the inclusion and exclusion criteria will be selected for inclusion.

   4.2 Treatment plan selection: A. Patients with T2N0 pyriform sinus cancer and posterior hypopharyngeal wall cancer will enter surgery directly; B. Patients with T2N1-3 or T3/N0-3 hypopharyngeal cancer will undergo surgery according to the patient's preference: a. 2-3 cycles of neoadjuvant chemotherapy (NAC) (PF regimen as usually) before entering re-evaluation. Immunotherapy with PD-1 monoclonal antibody is recommended for those with PD-L1 immunohistochemistry CPS score > 1; b. Those who refuse NAC directly go for surgery or radiotherapy (RT). After 2 cycles of induction therapy, laryngoscopy and MR/CT examination were performed and re-evaluated. According to the response evaluation criteria in solid tumor (RECIST) version 1.1, the efficacy of chemotherapy was evaluated as complete response (CR), partial response (PR), stable disease (SD) or progression disease (PD). According to the patient willingness to undergo surgery + postoperative RT, or CRT.

   4.3 Surgical methods: The patient undergoes tracheotomy under general anesthesia, and after neck dissection on the ipsilateral or both sides, incision is made from the front midline of the neck to expose the larynx. In T2 cases, the piriform sinus or posterior hypopharynx on the affected side is performed according to the tumor extent. Piriform sinus resection ± vertical hemi-lararyngectomy was performed in T3 tumor. The SMAIF was harvested and inserted through the lateral space of the patient's strap muscle to repair the defect of the ipsilateral hemi-larynx and hypopharynx.
5. Outcomes and Measures:

   5.1 Laryngeal function evaluation: laryngeal function evaluation is performed before surgery and 2 weeks, 1 month, 3 months, and 6 months after surgery. For patients who undergo radical radiotherapy, the laryngeal function evaluation is performed at 2 weeks, 1 month, 3 months, and 6 months after the end of treatment. Laryngeal function assessment includes: A. Voice function: stroboscopic laryngoscope/fiberoptic laryngoscope, voice aerodynamic examination, VHI-10 scale and GRBAS score; B. Respiratory function: postoperative tracheal tube removal time and removal rate; C. Swallowing function: Kubota test, gastric tube removal time, gastric tube removal rate.

   5.2 Follow-up and survival: In the first 2 years after surgery, outpatient follow-up visits will be performed every 3 months, laryngoscopy will be performed routinely, and neck MR or CT will be reviewed every 6 months. From the 3rd to 5th year after surgery, outpatient follow-up visits were performed every 6 months, laryngoscopy was performed routinely, and neck MR or CT was reviewed every 1 year. Overall survival (OS), disease-free survival (DFS), disease-specific survival (DSS) will be recorded routinely.
6. Ethical Considerations:

   This study complied with the 'Criterions for the Quality Control of Clinical Trial of drugs' and the "Management Measures for Investigator-Initiated Clinical Research in Medical and Health Institutions" (Trial) and the Declaration of Helsinki. Before the start of the trial, the study can only be carried out after the protocol has been approved by the ethics committee of our hospital. During the research process, if the protocol must be revised, the revised protocol must be resubmitted to the ethics committee for review, and the researcher must wait until the ethics committee agrees before implementing the new protocol.

   Each enrolled patient must sign an informed consent form. A copy of the informed consent form and the contact information of the researcher and ethics committee must be provided to the subject. This study will collect the clinical data and personal information of the research subjects for scientific research, and will involve the privacy rights of the patients. Participants and data analysts in this study have signed confidentiality contracts and will not disclose patient personal information and disease-related information to any individuals or institutions unrelated to this study. The collected patient data is managed in a unified manner to prevent the leakage of personal privacy.
7. Statistical Analysis:

7.1 Simple size estimation: the main indicator of this study is the laryngeal preservation rate (LPR). According to previous literature reports, the LPR of hypopharyngeal cancer rescetion is about 60%. According to a small sample of submental flap repair for hypopharyngeal cancer reported by He et al., the LPR is 88%. In this study, the LPR was set at 80%, and the selection ratio of T2:T3 is 1:2. According to the increase in the throat preservation rate from 60% to 80%, the type I error is one-sided 0.05, and the power is 0.8. Using the sample size calculation software PASS 15.0, the calculation requires 36 cases. Considering the dropout rate of 10%, a total of 40 cases are needed.

7.2 Statistical analyzes will be performed using SPSS software version 25 or higher. Continuous variables will be summarized using descriptive statistics (number of cases, mean, standard deviation, median, minimum, and maximum). Categorical variables were reported as frequencies and percentages. The time-to-event variable will be summarized using event and censoring frequencies, time-to-time quartiles.

For LPR, point estimates were performed and two-sided 95% confidence intervals were estimated using the Clopper-Pearson exact probability method.

Survival was summarized descriptively using the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

* T2-T3 hypopharyngeal squamous cell carcinoma located in the piriform sinus or posterior hypopharyngeal wall cancer;
* The contralateral hemilarynx is mobile;
* the Eastern Cooperative Oncology Group (ECOG) performance status (PS) score was 0 or 1;
* Without a history of radiotherapy.

Exclusion Criteria:

* Invasion into the cricoid cartilage and unable to reserve the larynx；
* Pulmonary insufficiency, FEV1/FVC<50%;
* Unresctable neck diseases including carotid artery envoloped or tumor penetration to the prevertebral fascia or mediastinum;
* Heart insufficincy whice intolerate to general anesthesia;
* With distant metastasis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2028-02-16 (Estimated); Study Completion 2030-02-16 (Estimated)

PRIMARY OUTCOMES:
The survival of submental artery island flap | one month after the end of the treatment
  The survival rate of submental artery island flap (SMAIF)
The recovery of laryngeal function | one month after the end of the treatment
  the removal of nasogastric tube and tracheal tube

SECONDARY OUTCOMES:
Overall survival of patients underwent the treatment with SMAIF reconstruction. | 2-year and 5-year after the initiation of treatment
  Overall survival
Disease-free survival of patients underwent the treatment with SMAIF reconstruction. | 2-year and 5-year after the initiation of treatment
  Disease-free survival
Local control rate of patients underwent the treatment with SMAIF reconstruction. | 2-year and 5-year after the initiation of treatment
  Local control rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Huang, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jang JY, Kim EH, Cho J, Jung JH, Oh D, Ahn YC, Son YI, Jeong HS. Comparison of Oncological and Functional Outcomes between Initial Surgical versus Non-Surgical Treatments for Hypopharyngeal Cancer. Ann Surg Oncol. 2016 Jun;23(6):2054-61. doi: 10.1245/s10434-016-5088-4. Epub 2016 Jan 19. PMID 26786092
- [Background] Martin D, Pascal JF, Baudet J, Mondie JM, Farhat JB, Athoum A, Le Gaillard P, Peri G. The submental island flap: a new donor site. Anatomy and clinical applications as a free or pedicled flap. Plast Reconstr Surg. 1993 Oct;92(5):867-73. PMID 8415968
- [Background] Chen R, Cai Q, Lin P, Liang F, Han P, Zhang L, Song P, Zhang T, Huang X. Role of immune-inflamed phenotype in the prognosis of hypopharyngeal carcinoma following primary surgery. Head Neck. 2023 Jan;45(1):126-134. doi: 10.1002/hed.27218. Epub 2022 Oct 12. PMID 36222335
- [Result] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Result] Garneau JC, Bakst RL, Miles BA. Hypopharyngeal cancer: A state of the art review. Oral Oncol. 2018 Nov;86:244-250. doi: 10.1016/j.oraloncology.2018.09.025. Epub 2018 Oct 4. PMID 30409307
- [Result] Habib A. Management of advanced hypopharyngeal carcinoma: systematic review of survival following surgical and non-surgical treatments. J Laryngol Otol. 2018 May;132(5):385-400. doi: 10.1017/S0022215118000555. PMID 29891019
- [Result] Eckel HE, Bradley PJ. Treatment Options for Hypopharyngeal Cancer. Adv Otorhinolaryngol. 2019;83:47-53. doi: 10.1159/000492308. Epub 2019 Feb 12. PMID 30943512
- [Result] Cai Q, Liang F, Huang X, Han P, Pan Y, Zheng Y. Hypopharynx and larynx defect repair after resection for pyriform fossa cancer with a platysma skin flap. Otolaryngol Head Neck Surg. 2015 Feb;152(2):374-6. doi: 10.1177/0194599814559508. Epub 2014 Nov 26. PMID 25428776
- [Result] Chen L, Si Y, Lin P, Guan Z, Zhu W, Liang H, Cai Q. Surgical treatment of T2-3 posterior hypopharyngeal carcinoma with preservation of laryngeal function. Acta Otolaryngol. 2021 Sep;141(9):851-856. doi: 10.1080/00016489.2021.1965211. Epub 2021 Aug 30. PMID 34459710
- [Result] Pang W, Zhang A, Lu C, Tian J, Li WX, Wang Z, Dong Y, Yuan S, Niu Z, Zhu Y, Quraishi MS, Liu L. Design and application of submental island flap to reconstruct non-circumferential defect after hypopharyngeal carcinoma resection: a prospective study of 27 cases. Acta Otolaryngol. 2020 Dec;140(12):1036-1042. doi: 10.1080/00016489.2020.1804614. Epub 2020 Aug 18. PMID 32808843